CLINICAL TRIAL: NCT02248051
Title: An Open-Label, Non-Randomized Study of Safety, Tolerability and Pharmacokinetics of Intravenous CXA-10 Emulsion in Subjects With Stage 3 and 4 Chronic Kidney Injury
Brief Title: Open-Label Safety, Tolerability, PK Study of IV CXA-10 Emulsion in Subjects in Chronic Kidney Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Complexa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXA-10-002
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2016-05

CONDITIONS: Acute Kidney Injury (Nontraumatic)
MeSH Terms: conditions — Acute Kidney Injury | interventions — CXA-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CXA-10 (Experimental)
  Interventions: Drug: CXA-10

INTERVENTIONS:
Drug: CXA-10 — CXA-10 Injectable Emulsion is a sterile emulsion containing CXA-10 in a formulation containing soybean oil, medium chain triglycerides oil, egg phospholipids, sucrose, and disodium EDTA. CXA-10 Injectable Emulsion will be administered intravenously. The active emulsion will be diluted in a vehicle emulsion.

SUMMARY:
The main purpose of this trial is to demonstrate the safety, tolerability and pharmacokinetics (PK) of CXA-10, at potentially therapeutic doses, in the target patient population comprised of subjects with Stage 3 and 4 chronic kidney injury (CKI). In addition, associated pharmacodynamic (PD) effects of CXA-10 will be investigated.

DETAILED DESCRIPTION:
This will be a multi-center, open-label study, single-dose study with CXA-10 in subjects with CKI. At total of 12 subjects will be enrolled into two equal groups according to their baseline estimated glomerular filtration rate (eGFR: 15 - 39 or 40 - 59 mL/min/1.73m2). All subjects will receive a single dose infusion of CXA-10 emulsion. Since this is the first administration of CXA-10 to a non-healthy volunteer population, a conservative approach is being taken to ensure safety. Thus, the first 2 subjects from each group will be dosed at one dose level below the highest safe dose level administered in the FIH study. If this dose is found to be safe in this specific subject population, the remainder of the 4 subjects in each group will receive the highest safe dose from the FIH study; otherwise, the remainder will receive the initial dose. The doses administered in this study will not exceed the highest exposures achieved in the FIH study, and doses may need to be adjusted to lower levels, based on further evaluation of current pharmacokinetic data, to ensure the appropriate the exposure level. Safety, PK and PD assessments will be conducted over approximately 18 days following each dosing session. There will be a follow-up visit approximately 1 week after dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of non-child bearing potential 18 to 70 years of age (inclusive).
2. Moderate to severe CKI (equivalent to National Kidney Foundation Kidney Disease Outcomes Quality Initiative [NKF KDOQI] Stage 3 or 4, not receiving dialysis) as determined by estimated glomerular filtration rate (eGFR) greater than or equal to 15 and less than 60 mL/min/1.73 m2 (according to the creatinine-cystatin C equation) within less than or equal to 3 months prior to the screening visit. Cause of the CKI should be recorded where possible.
3. Body mass index (BMI) between 18 and 40 kg/m2 (inclusive)
4. Subjects must have resting heart rates (HR) greater than or equal to 50 beats per minute at baseline
5. QTcF interval (Fredericia's correction factor) of the baseline ECG must be less than or equal to 450 msec for males and less than or equal to 470 msec for females at screening and predose. Subjects with any other clinically relevant ECG parameter abnormality (e.g., PR interval, QRS deviation) or any clinically significant ECG abnormality will be excluded from the study. Subjects with a history of congenital long QT syndrome or short QT syndrome in the subject or in the subject's family will be excluded from the study.
6. Adequate bilateral venous access to allow for dose infusions and blood sampling
7. Ability to comprehend and comply with procedures
8. Agree to commit to participate in the current protocol
9. Provide written informed consent prior to any study procedure being performed

Exclusion Criteria:

1. Female subjects who are pregnant or lactating or who are trying to conceive
2. Female subjects with a positive serum β-human chorionic gonadotropin (β-hCG) test at screening or Day -1 for any dosing day
3. History of renal transplantation
4. History of acute dialysis or acute kidney injury within 12 wks prior to screening and dosing
5. Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) 3.0X upper limit of normal (ULN), gamma-glutamyl transferase (GGT) greater than 3X ULN, and total bilirubin greater than 2X ULN. If all liver function tests (LFTs) are within normal limits (WNL) and total bilirubin is elevated, examination of direct and indirect bilirubin may be conducted. Subjects with indirect total bilirubin up to 3X ULN are presumed to have Gilbert's syndrome and may be enrolled if all other LFTs are WNL.
6. Presence of signs and symptoms of uremia
7. Past history of pancreatitis
8. History of documented hypersensitivity reaction to eggs or egg products (as the vehicle contains egg phospholipids)
9. History of documented hypersensitivity reaction to soy or soy products (as vehicle contains soy bean oil)
10. Uncontrolled diabetes with HbA1c > 9 percent or subjects with frequent hypoglycemic attacks
11. Active cardiovascular disease within 12 weeks of dosing, including unstable angina, myocardial infarction, coronary artery bypass or percutaneous transluminal angioplasty/stent, cerebrovascular accident including transient ischemic attack, any history of syncope, dizziness, cardiac arrhythmias, cardiac arrest, pacemakers, cardioversion, and clinical diagnosis of severe obstructive valvular heart disease or severe hypertrophic cardiomyopathy
12. Current diagnosis of Class 3 or 4 New York Heart Association (NYHA) congestive heart failure.
13. Uncontrolled hypertension with sitting blood pressure greater than 160 mmHg systolic and or greater than 100 mmHg diastolic after 5 minutes rest (feet on floor, arm held at level of heart) at the screening visit
14. Resting heart rate greater than or equal to 100 beats per minute (BPM) after 5 minutes rest (as above) at the screening visit
15. Any abnormalities on 12-lead ECG, as deemed by the investigator and/or medical monitor, at screening
16. Any clinically significant murmurs evident on auscultation of the heart (including evidence of mitral valve prolapse)
17. History of smoking or use of nicotine-containing products in excess of approximately a pack per day (estimated at 20 cigarettes per day) or equivalent within the past 2 weeks
18. History of drug abuse or dependence within 6 months of the study
19. History of regular alcohol consumption within 6 months of the study, defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits.
20. A positive drug screen for drugs of abuse, including alcohol at the screening visit or at entry to the clinic
21. Treatment with any investigational drug within 30 days or 5 half-lives prior to the beginning of the screening period (this includes investigational formulations of marketed products, inhaled and topical drugs)
22. Blood collection of greater than 500 mL within 56 days prior to screening
23. Seropositive for human immunodeficiency virus (HIV) at screening
24. Positive for Hepatitis B virus surface antigen (HBsAg) or positive Hepatitis C virus antibody (HCV Ab) at screening
25. Any other condition and/or situation that causes the Investigator to deem a subject unsuitable for the study (e.g., due to expected study medication non compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study related procedures)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Serious and Non-Serious Adverse Events | First day of dosing through 30 days
  Safety assessments will be performed prior to, during, and after dosing including a visit on Day 18

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Jasper Clinical Research & Development, Inc., Kalamazoo, Michigan

IPD SHARING:
Plan to Share IPD: No